CLINICAL TRIAL: NCT02529735
Title: Etude Prospective Observationnelle Multicentrique Sur Volontaires Sains Des VALeurs de Pression Artérielle mesurées Sur Trois Sites alteRnAtIfS Des Membres inférieurs cOmparées au Site de référence
Brief Title: Study on Pressure Values Measured on Three Alternative Sites of the Lower Limbs Compared to the Arm
Acronym: VALPARAISO
Status: Available | Type: Expanded Access
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Principal Investigator, Steven Lagadec, Principal Investigator, Centre Hospitalier Sud Francilien
Other Study IDs: CHSFrancilien
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Blood Pressure
Keywords: blood pressure; alternative measure

INTERVENTIONS:
Other: efficiency study — Blood pressure values measured for comparative lower limb and arm

SUMMARY:
Non-invasive measurement of blood pressure is an instrument governed nursing routine care. The use of an automated oscillometric cuff is a common technique and validated if this is done on the arm with a suitable cuff, positioned opposite the brachial artery and up to the right atrium (the brachial site) . If cons-indication to use the brachial site, measurements are frequently performed at the ankle, calf or thigh. Among the blood pressure values measured on the 3 sites of the lower limb (thigh, calf or ankle), it may be a specific property of which the observed values are closest to the reference values (brachial).

The objective of this study is to measure the non-invasive blood pressure values at three sites of the lower limb, to compare the reference value to determine which alternative site should be preferred when the reference measurement is not feasible .

We want to determine the alternative site to obtain values as close as the measured values of the reference site. The three study sites are the thigh, calf and ankle. The reference site recommended for monitoring non-invasive blood pressureis the arm.

It is also assessing the impact of certain parameters on the primary endpoint:

* Physiological parameters: gender, weight, height, age, systolic blood pressure reference, listed measures.
* A parameter related to measurement: discomfort felt when the blood pressure outlet.
* Exposure setting: smoking.

DETAILED DESCRIPTION:
Primary Outcome: The difference in systolic blood pressure, diastolic and mean simultaneously measured in the arm and each of the three sites in the lower limb.

Secondary endpoints: The difference in systolic blood pressure, diastolic and mean simultaneously measured in the arm and each of the three sites in the lower limb in the following subgroups:

* Male / Female
* BMI <25 / BMI> 25
* Size < 160 cm / size [160-169] cm / size [170-180] cm / size [181-190] cm / size ≥ 191 cm
* Age <25 years / age ≥ 25 years
* Systolic Blood Pressure value (SAP) the reference site <100 mmHg / 100 mmHg and ≥ NOT value of the reference site <140 mmHg / ≥ 140 mmHg
* Visual Analog Scale of discomfort ≤ 4/10 /> 4/10
* Hemibody studied Right / Left
* Smoking / No Smoking

Discomfort level depending on the measurement site of blood pressure in the general population.

* Discomfort level for each measurement of blood pressure site in each of the following subgroups:
* Male / Female - BMI <25 / BMI> 25
* size <160 cm / size [160-169] cm / size [170 -180] cm / size [181-190] cm / size ≥ 191 cm - Age <25 / age ≥ 25 years
* blood pressure value (SAP) reference site <100 mmHg / 100 mmHg and ≥ NOT Value reference site <140 mmHg / ≥ 140 mmHg
* hemibody studied Right / Left
* Smoking / No Smoking

Methodology:

Experimental design:

This is an observational study, prospective, multicenter, comparative on healthy volunteers, each individual is his own witness. Reports of non-invasive blood pressure values of 3 different sites of the lower limbs, compared to a reference value. For each individual, the side which will be carried out blood pressure measurements will be drawn. After 5 minutes rest in the supine position, it will be realized the measurement of blood pressure non-invasively systolic, mean and diastolic 2 automated oscillometric measuring devices identical and calibrated simultaneously the arm and thigh ipsilateral / arm and calf ipsilateral / arm and the ipsilateral ankle.

Each measurement is repeated once after 1 minute.

Statistical analysis:

Systolic, mean and diastolic pressures are analyzed separately, and expressed by their average with standard deviation and 95% confidence intervals. The concordance of BP measurements between the arm and each of three sites in the lower limb was analyzed by the method Bland and Altman, calculating the average difference, its approval limits, as well as the confidence interval 95 % upper and lower limits of approval subject to a Gaussian distribution of the difference between the measurements.

The search for the best AP measurement site to the lower member is made by comparing the differences between each of the three sites and the reference site, for a global test (variance analysis or test Friedmann according to the distribution of differences), then by comparisons with 2-2 adjusting the p-value.

The chosen site is one for which this difference is significantly weaker. All tests are conducted bilaterally with a risk of first species set at 5%. In an earlier study, the largest variance found regarding the difference in systolic BP between calf and arm.

Based on the most pessimistic scenario (s = 12.76) to highlight a difference of 5 mm Hg with an alpha risk of 5% and a power of 90% and taking into account the multiple comparisons considered, 176 patients necessary.

Total duration of study: 27 months Period of inclusion: 24 months Duration of participation for voluntary: 30 minutes Number of participating centers: 8 centers

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over, without upper age limit
* Recipient of a social protection scheme or entitled
* Signature of informed consent

Exclusion Criteria:

* During Pregnancy
* known disease
* current treatment
* cardiovascular history
* Skin lesions in relation to the measurement sites
* Special anatomically incompatible with blood pressure measurements
* No one opposing the use of their data
* Participation in a trial Ongoing clinical
* Person who participated in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lagadec, RN, Study Director — Centre Hospitalier Sud Francilien
Locations (8):
- France (8):
  - Sud Francilien Nursing School, Corbeil-Essonnes
  - Perray-Vaucluse Nursing School, Épinay-sur-Orge
  - Nursing Scool Barthelemy Durand, Étampes
  - SSSM of Essonne SDIS91, Évry
  - Nursing School of Longjumeau, Longjumeau
  - Nursing School Tenon, Paris
  - Nursing School Rambouillet, Rambouillet
  - Nursing School Foch, Suresnes

REFERENCES:
- [Result] Chatterjee A, DePriest K, Blair R, Bowton D, Chin R. Results of a survey of blood pressure monitoring by intensivists in critically ill patients: a preliminary study. Crit Care Med. 2010 Dec;38(12):2335-8. doi: 10.1097/CCM.0b013e3181fa057f. PMID 20890190
- [Result] Block FE, Schulte GT. Ankle blood pressure measurement, an acceptable alternative to arm measurements. Int J Clin Monit Comput. 1996 Aug;13(3):167-71. doi: 10.1023/a:1016997232542. PMID 8912031
- [Result] Sanghera S, North A, Abernethy S, Wrench I. Arm and ankle blood pressure during caesarean section. Int J Obstet Anesth. 2006 Jan;15(1):24-7. doi: 10.1016/j.ijoa.2005.04.016. Epub 2005 Oct 26. PMID 16256340
- [Result] Moore C, Dobson A, Kinagi M, Dillon B. Comparison of blood pressure measured at the arm, ankle and calf. Anaesthesia. 2008 Dec;63(12):1327-31. doi: 10.1111/j.1365-2044.2008.05633.x. PMID 19032301
- [Result] Lakhal K, Macq C, Ehrmann S, Boulain T, Capdevila X. Noninvasive monitoring of blood pressure in the critically ill: reliability according to the cuff site (arm, thigh, or ankle). Crit Care Med. 2012 Apr;40(4):1207-13. doi: 10.1097/CCM.0b013e31823dae42. PMID 22425818